CLINICAL TRIAL: NCT06158425
Title: Distribution of Coronal Plane Alignment of the Knee Classification in Chinese Osteoarthritic as Well as Healthy Population
Brief Title: Constitutional Alignment in Osteoarthritic and Healthy Chinese
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: FirstJilinUQX
Record Dates: First submitted 2023-11-26; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OA group: Data for consecutive OA patients with knee pain who underwent primary TKA by one senior surgeon between August 2021 and July 2023 at a single institution were analyzed retrospectively. A total of 273 patients underwent long-leg radiographs. The following 27 patients were excluded from this study: prior total hip arthroplasty, 2; obvious bony deficiency of the femur or tibia, 10; simultaneous flexion of the knee and rotation of the leg on radiographs, 15. CPAK distribution of the remaining 246 cases(unilateral, 15; bilateral, 231; totally 477 knees) was examined.
  Interventions: Radiation: long-leg radiograph
- healthy group: Data for consecutive visitors at outpatient clinic who underwent long-leg radiographs but without any sign of cartilage degeneration or medical history of low extremity between January 2023 and July 2023 at the same institution were analyzed retrospectively. A total of 136 visitors were recruited. The following 18 visitors were excluded from this study: extra-articular deformity of the femur or tibia, 15; simultaneous flexion of the knee and rotation of the leg on radiographs, 13; poor quality image, 1. CPAK distribution of the remaining 107 cases(214 knees) was examined.
  Interventions: Radiation: long-leg radiograph

INTERVENTIONS:
Radiation: long-leg radiograph — A flat-panel digital radiography(DR) equipment (Siemens DR AXIOM Aristos AX/VX) was used to capture full-length bipedal lower extremities in a standing position. The technician moved the detector from top to bottom, capturing four parts: the bilateral hip joints, femur, tibia and fibula and ankle joint. The exposure parameters for each part were as follows: 1st exposure - 85kV, 75mAs; 2nd exposure - 80kV, 50mAs; 3rd exposure - 75kV, 40mAs; 4th exposure - 68kV, 20mAs. The distance from the source (kv-kg) was 300cm, and the field of view was 43.18cm x 43.18cm. All 4 X-rays were stitched using the Siemens DR Station.

SUMMARY:
coronal plane alignment of the knee(CPAK) distribution of 246 cases(477 knees) of OA patients and 107 cases(214 knees) of healthy people were examined on long-leg radiographs retrospectively. Radiological measurements and CPAK classification on different Kellgren- Lawrence(K-L) Grade in patients with unilateral total knee arthroplasty(TKA) were compared. Clinical outcomes of CPAK type I patients performed by mechanical alignment(MA) and restricted kinematic alignment(rKA) during TKA were examined. ML algorithm including K nearest neighbors (KNN), random forest(RF), artificial neural networks (ANN), logistic regression(LR) and gradient boosting (GBDT) were established, the dependent variable was set as whether the constitutional phenotype of an arthritic knee classified as type I was type I.

DETAILED DESCRIPTION:
Study groups and design OA group Data for consecutive OA patients with knee pain who underwent primary TKA by one senior surgeon between August 2021 and July 2023 at a single institution were analyzed retrospectively. A total of 273 patients underwent long-leg radiographs. The following 27 patients were excluded from this study: prior total hip arthroplasty, 2; obvious bony deficiency of the femur or tibia, 10; simultaneous flexion of the knee and rotation of the leg on radiographs, 15. CPAK distribution of the remaining 246 cases(unilateral, 15; bilateral, 231; totally 477 knees) was examined.

healthy group Data for consecutive visitors at outpatient clinic who underwent long-leg radiographs but without any sign of cartilage degeneration or medical history of low extremity between January 2023 and July 2023 at the same institution were analyzed retrospectively. A total of 136 visitors were recruited. The following 18 visitors were excluded from this study: extra-articular deformity of the femur or tibia, 15; simultaneous flexion of the knee and rotation of the leg on radiographs, 13; poor quality image, 1. CPAK distribution of the remaining 107 cases(214 knees) was examined.

Radiological measurements All participants underwent standard digital long leg radiographs. The mechanical axis of the femur was marked from the centre of the femoral head to the centre of the knee. The centre of the head was marked using the concentric-circle method to identify the centre. The centre of the ankle was marked as the point on the talar dome at mid-width. The mHKA angle was the angle subtended by the mechanical axes of the femur and tibia. The LDFA was defined as the lateral angle formed between the femoral mechanical axis and the joint line of the distal femur. The MPTA was defined as the medical angle formed between the tibial mechanical axis and the joint line of the proximal tibia. Joint line convergence angle(JLCA) was the angle formed between joint orientation lines on opposite sides of the same joint[17]. All measurements were carried out by an orthopaedic fellow. A senior author undertook a subgroup analysis of 60 knees in OA group and repeated at one- week intervals to assess for inter- and intra- observer agreement.

CPAK classification of OA and healthy group aHKA was calculated based on the following formula: aHKA=MPTA-LDFA. JLO was calculated by the formula: JLO=MPTA+LDFA. With aHKA and JLO measured, patients can be matched to 9 possible CPAK alignment groups. The mean aHKA and JLO of the two groups were rounded to the nearest whole number for final allocation to a CPAK Class. CPAK limits for the definition of neutral knees was an aHKA of 0 ± 2 degrees. CPAK boundaries for a neutral JLO were defined as 180 ± 3 degrees, varus aHKA less than-2 degrees and a valgus aHKA more than+2 degrees. An apex distal JLO was less than 177°, while an apex proximal JLO was greater than 183°[9]. The OA and healthy group were categorized according to the CPAK classification, and their distribution were investigated.

ELIGIBILITY:
Inclusion Criteria:

- OA group: Data for consecutive OA patients with knee pain who underwent primary TKA by one senior surgeon between August 2021 and July 2023 at a single institution were analyzed retrospectively.

Healthy group: Data for consecutive visitors at outpatient clinic who underwent long-leg radiographs but without any sign of cartilage degeneration or medical history of low extremity between January 2023 and July 2023 at the same institution were analyzed retrospectively.

Exclusion Criteria:

- OA group: prior total hip arthroplasty; obvious bony deficiency of the femur or tibia, simultaneous flexion of the knee and rotation of the leg on radiographs Healthy group: extra-articular deformity of the femur or tibia; simultaneous flexion of the knee and rotation of the leg on radiographs; poor quality image

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: OA group: consecutive OA patients with knee pain who underwent primary TKA Healthy group: consecutive visitors at outpatient clinic who underwent long-leg radiographs but without any sign of cartilage degeneration or medical history of low extremity
Sampling Method: Non-Probability Sample
Enrollment: 353 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-06 (Estimated)

PRIMARY OUTCOMES:
CPAK distribution | before surgery
  distribution of coronal plane alignment of the knee classification

CONTACTS AND LOCATIONS:
Overall Officials: Bin Liu, Study Chair — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao YH, Qi YM, Huang PH, Zhao XY, Qi X. Joint line convergence angle should be considered when constitutional alignment is predicted based on arithmetic hip-knee-ankle angle: a retrospective cross-sectional observational study. Int J Surg. 2025 Jan 1;111(1):1624-1628. doi: 10.1097/JS9.0000000000002097. PMID 39361874
- [Derived] Gao YH, Qi YM, Huang PH, Zhao XY, Qi X. Distribution of coronal plane alignment of the knee classification in Chinese osteoarthritic and healthy population: a retrospective cross-sectional observational study. Int J Surg. 2024 May 1;110(5):2583-2592. doi: 10.1097/JS9.0000000000001178. PMID 38349219